CLINICAL TRIAL: NCT00582413
Title: Prospective Evaluation of Quality of Life and Development of Measures in Patients With Cancer of the Oral Cavity
Brief Title: Quality of Life and Development of Measures in Patients With Cancer of the Oral Cavity
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Monash University (Other)
Responsible Party: Sponsor
Other Study IDs: 04-137
Record Dates: First submitted 2007-12-21; First posted 2007-12-28 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Cancer of the Oral Cavity
Keywords: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: Patients who have been diagnosed with Carcinoma of the oral cavity
  Interventions: Behavioral: questionnaires

INTERVENTIONS:
Behavioral: questionnaires — Patient will fill out questionnaires, initial clinic visit, first post-surgery clinic evaluation and 3, 6, 12, 18 and 24 months following completion of all therapy.

SUMMARY:
The purpose of this study is to learn more about the quality of life and emotional changes that patients experience during their treatment for cancer of the mouth. We want to learn more about the emotional and quality of life problems that occur during and after treatment. This will help us better understand these complex issues and improve treatment.

DETAILED DESCRIPTION:
The objectives of this project are to prospectively assess quality of life (QOL) and psychosocial adaptation in patients undergoing treatment for carcinoma of the oral cavity, including squamous cell carcinoma of the oral cavity (SCCOC) and to validate new instruments (shame & stigma, demoralization) that will guide quality of life assessment of patients with cancer of the oral cavity. We will utilize modifications of previously described and validated questionnaires that will be administered to eligible patients before the start of their therapy and at several predefined time points during the post-therapy period. This prospective longitudinal assessment will allow us to study the impact of patient demographic, tumor, treatment and lifestyle related variables on the quality of life of patients treated for oral cavity cancer.

ELIGIBILITY:
Inclusion Criteria:

PATIENT INCLUSION CRITERIA FOR THE LONDITUDINAL STUDY:

* Carcinoma of the oral cavity including one or more of the following anatomic sub-sites: Anterior 2/3rds of the tongue, the floor of the mouth, the upper and lower gums, buccal mucosa, retromolar trigone, hard palate and minor salivary glands.
* Surgically resectable disease in the oral cavity and the neck.
* Patients with prior cancers other than Head and Neck cancers who are currently in remission, have no evidence of disease and are not undergoing any active chemotherapy or radiation therapy.

Exclusion Criteria:

EXCLUSION FOR THE LONDITUDINAL STUDY:

* Primary tumor of the lips (these are skin cancers).
* Surgical treatment excluding diagnostic biopsy of the primary site or biopsy of neck node/s prior to referral to MSKCC.
* Surgically unresectable disease in the neck; including carotid encasement, massive dermal infiltration, and other clinical and radiographic findings which would preclude surgically resectable nodal disease in the neck, prior to initiation of treatment.
* Evidence of distant metastases by clinical or radiographic examination.
* Patients with more than one simultaneous primary tumor.
* Patient unable to read or comprehend the content of the questionnaires due to language barriers or psychiatric disorders.

PATIENT INCLUSION CRITERIA FOR THE CROSS-SECTIONAL STUDY:

* Upper aerodigestive squamous cell carcinoma, including the oropharynx, hypopharynx and larynx - newly diagnosed or recurrent cancers.
* Newly diagnosed and recurrent carcinoma of the oral cavity including one or more of the following anatomic sub-sites: Anterior 2/3rds of the tongue, the floor of the mouth, the upper and lower gums, buccal mucosa, retromolar trigone, hard palate and minor salivary glands.

EXCLUSION CRITERIA FOR THE CROSS-SECTIONAL STUDY:

* Primary tumor of the lips (these are skin cancers).
* Patient unable to read or comprehend the content of the questionnaires due to language barriers or psychiatric disorders.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients seen on the Head and Neck Surgery Service, Radiation Oncology Service, Medical Oncology Service and Dental Service.
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2004-12; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
is to assess quality of life and psychosocial adaptation in patients undergoing treatment for cancer of the oral cavity so that we can develop empirically-informed interventions to improve the adaptation of these patients. | conclusion of study

SECONDARY OUTCOMES:
Validate two new measures of psychosocial adjustment in patients treated for cancer of the oral cavity and upper aerodigestive SCC: The Shame and Stigma in Head and Neck Cancer Scale and the Demoralization Scale | conclusion of study
Assess patterns of tobacco and/or alcohol use in cancer of the oral cavity survivors. | conclusion of the study
Assess the impact of lifestyle and socio-economic issues on post-therapy quality of life. | conclusion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Snehal Patel, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org